CLINICAL TRIAL: NCT03093493
Title: Determine the Causative Genetic Variations in Patients With Ehlers-Danlos Syndrome
Brief Title: Genetics of Ehlers-Danlos Syndrome
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: H-36286
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Genetics Syndrome; Ehlers-Danlos Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Ehlers-Danlos Syndrome | interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood and saliva for DNA extraction to use in genetic testing of children and adults with EDS and their relatives will be collected. Medical records from other institutions and notes from visits in Dr. Holick's clinic will be reviewed to obtain the following information: previous diagnosis at other institutions, age, clinical signs and symptoms of EDS, Joints Hypermobility Syndrome (JHS), other metabolic or genetic disorders and laboratory results, radiology reports and images, and genetic testing that support these diagnoses. Subjects' peripheral vein blood, saliva and pictures will be taken. A clinical evaluation will be performed to document clinical signs for EDS. No clinical interventions will be performed. No patients' identifiers will be reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EDS patients: Medical records from other institutions and clinical notes for visits in Dr. Holick's clinic will be reviewed to obtain the following information: previous diagnosis at other institutions, age, clinical signs and symptoms of EDS, Joints Hypermobility Syndrome (JHS), and other metabolic or genetic disorders and laboratory results, radiology reports and images, and genetic testing that supports EDS diagnoses. Genotyping will be done.
  Interventions: Diagnostic Test: Genotyping
- EDS family members with or without EDS: Family members of EDS patients with or without EDS. Genotyping will be done.
  Interventions: Diagnostic Test: Genotyping

INTERVENTIONS:
Diagnostic Test: Genotyping — Genotyping by next generation sequencing

SUMMARY:
We are planning to collected blood and saliva for DNA extraction to use for genetic testing of children and adults with EDS and their relatives. Medical records from other institutions and clinical notes for visits in Dr. Holick's clinic will be reviewed to obtain the following information: previous diagnosis at other institutions, age, clinical signs and symptoms of EDS, Joints Hypermobility Syndrome (JHS), , and other metabolic or genetic disorders and laboratory results, radiology reports and images, and genetic testing that supports these diagnoses. Subjects' peripheral vein blood and saliva will be taken. No clinical intervention/randomizations will be performed. No patients' identifiers will be reported.

In this pilot study genomic DNA will be extracted and will be used for genotyping as sequencing in 30 EDS patients and their 30 relatives with or without EDS to compare genetic variations between them. After validation by Sanger sequencing for these variations, we plan to prepare a genetic panel for EDS. After all validation testing, we plan to evaluate the saliva DNA in a similar manner and compare the results with those obtained from the DNA from the blood sample. The purpose is that if they are comparable, we will be able to use saliva in place of blood as it easier method for accessing a person's DNA. This will be especially helpful for evaluating infants or those patients who prefer not to have a blood sample drawn. NOTE: Results of this study will not be disclosed to subjects.

DETAILED DESCRIPTION:
Ehlers-Danlos Syndrome (EDS) is a genetic disease that affects collagen synthesis and structure resulting in multisystem connective tissue involvement with twelve different subtypes. The clinical manifestations of EDS include skin hyperextensibility, skin fragility, joint hypermobility, muscle hypotonia, easy bruising, and mast cell hypersensitivity. We recently reported a cases series of EDS patients with different signs and symptoms. Most were evaluated along with their parents for evidence of acquired or inherited bone diseases. What is remarkable is that 93% of our cases at least one parent had clinically documented evidence for EDS a genetic disorder that compromises the structural integrity of the collagen/elastin matrix. Most of the parents were unaware they had this genetic disorder and the diagnosis was made for the first time in our clinic. Our previous study for reviewing patient's medical records was approved by the Boston University Medical Center's IRB. We have access to EDS patients from referrals and from Dr Holick's clinic. We plan to collect the blood and saliva samples from EDS patients and their relatives for this genetic study.

Genetic evaluation in limited number of our patients showed some causative variations. For example, one of our cases the patient was evaluated at an outside hospital for a causative variant in the COL5A1, COL5A2, FKBP14, and TNXB genes, which were negative, but she was found later to have a causative variant in serpin peptidase inhibitor, clade F, member 1 (SERPINF1) gene. A causative variation in SERPINF1 gene has been associated with osteogenesis imperfecta (OI) /EDS overlap syndrome and the mutation in this gene causes type VI OI.

The highly variable clinical presentation of patients with the hypermobility and clinical signs for EDS prompted an effort to classify patients with EDS into more homogeneous groups that can aid in diagnosis and management. This resulted in the establishment of 14 types (include 6 major types and 8 minor types). This classification acknowledges the presence of "others" including "unspecified" forms making it clear that the clinical and genetic heterogeneity of EDS could not be fully captured by that classification. Indeed, there have been numerous reports of patients with hereditary disorders of connective tissue, which have overlapping clinical manifestations of EDS, but do not meet the diagnostic criteria.

For decades, the genetic basis of heritable disorders of connective tissue had remained largely unknown. The rise of molecular genetics and its advances in next-generation sequencing has unlocked doors that continues to lead to major advances in understanding the causative genes for many genetic disorders.

Evaluation of subjects with these conditions often includes molecular testing which has important counseling, therapeutic and sometimes legal implications. An accurate molecular diagnosis can provide the basis for counseling regarding prognosis and reproductive options. Accurate genetic diagnosis has been shown to provide psychological benefits to patients and their families. In order to facilitate sequencing of multiple genes causing some of the common forms of these heritable conditions, we have designed this genetic study to obtain data for the genetic variations of EDS by next generation sequencing. The next generation sequencing panel may be of value in guiding future clinical pathways for genetic diagnosis in EDS. We plan to recruit EDS patients and their relatives for genetic testing. We also plan to submit a NIH grant for this purpose and provide required preliminary data through this pilot grant about genetic variation of EDS.

The primary objective is to compare genetic variations in EDS patients with their relatives. We expect to find some genetic variations that may explain clinical signs and symptoms in EDS patients.

Secondary objective is to provide a novel testing panel on a single diagnostic platform for EDS. After performing next generation sequencing, we plan to design a genetic panel for EDS.

A third objective will be to determine if saliva can be as good and reliable source of DNA for genetic testing as DNA obtained from blood.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults of any age

  * Both gender
  * Positive history of hypermobility or other related signs/symptoms of EDS these include among others a history of gastroparesis, orthostatic hypotension and easy bruising in EDS patient group.

Exclusion Criteria:

* Diagnosed as other metabolic or genetic disorders in EDS suspected subjects.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical records from other institutions and clinical notes for visits in Dr. Holick's clinic will be reviewed to obtain the following information: previous diagnosis at other institutions, age, clinical signs and symptoms of EDS, Joints Hypermobility Syndrome (JHS), , and other metabolic or genetic disorders and laboratory results, radiology reports and images, and genetic testing that supports EDS diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Causative genetic variations relation to EDS | one year
  Comparing genetic variations between EDS patients and their family memebers with or without EDS by next generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holick, MD PhD, Principal Investigator — Boston Univeristy
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No